CLINICAL TRIAL: NCT02932254
Title: Magnesium Sulfate Effect Following the Reversal of Neuromuscular Blockade Induced by Rocuronium With Sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Paulo Alipio Germano Filho, MD, MSc, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAGF02MG
Record Dates: First submitted 2016-07-25; First posted 2016-10-13 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Neuromuscular Blockade
Keywords: Physiological Effects of Drugs; Rocuronium; Sugammadex sodium; Magnesium; Neuromuscular block, antagonism
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium Sulfate (Active Comparator): 1. After anaesthesia induction and calibration of neuromuscular monitoring (acceleromyography) 0,6 mg/kg of rocuronium is given intravenously.
  2. After recovery of the neuromuscular block to a posttetanic count of 2 (deep neuromuscular block) or reappearance of 2 twitches of the train of four (moderate neuromuscular block), 4 mg/kg (deep neuromuscular block) or 2 mg/kg (moderate neuromuscular block) of sugammadex are given intravenously.
  3. INTERVENTION: After 90% of baseline T4 / T1, are injected intravenously magnesium sulfate 60 mg/kg over 10 minutes (100 mL solution).
  Interventions: Drug: Magnesium Sulfate
- Saline Solution (Placebo Comparator): 1. After anaesthesia induction and calibration of neuromuscular monitoring (acceleromyography) 0,6 mg/kg of rocuronium is given intravenously.
  2. After recovery of the neuromuscular block to a posttetanic count of 2 (deep neuromuscular block) or reappearance of 2 twitches of the train of four (moderate neuromuscular block), 4 mg/kg (deep neuromuscular block) or 2 mg/kg (moderate neuromuscular block) of sugammadex are given intravenously.
  3. INTERVENTION: After 90% of baseline T4 / T1, are injected intravenously 100 mL saline solution over 10 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Magnesium Sulfate — After 90% of baseline T4 / T1, are injected intravenously magnesium sulfate 60 mg/kg over 10 minutes (100 mL solution).
  Other Names: magnesium sulphate
  Arms: Magnesium Sulfate
Drug: Saline — After 90% of baseline T4 / T1, are injected intravenously saline solution over 10 minutes (100 mL solution).
  Other Names: NaCl 0,9%
  Arms: Saline Solution

SUMMARY:
The aim of this study is to evaluate the treatment effect of magnesium sulfate on the T4 / T1 ratio after reversal with sugammadex deep or moderate neuromuscular blockade induced by rocuronium.

DETAILED DESCRIPTION:
Sugammadex is a novel neuromuscular blocking reversal agent. Its mechanism of action is the encapsulation of rocuronium and vecuronium molecules. Numerous studies show a potential role of magnesium in reducing anesthetic requirements, sympathetic response to surgical trauma, antinociceptive action and neuroprotective effects. However, its use is limited because magnesium potentiates non-depolarizing neuromuscular blocking agents.

Primary outcome: evaluating the effect of treatment with magnesium sulfate the T4 / T1 ratio after reversal with sugammadex deep and moderate neuromuscular blockade induced by rocuronium.

Secondary outcome: evaluate the occurrence of severe respiratory events, the incidence of residual neuromuscular block in the post-anesthetic recovery room, evolution of T1 high, and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2
* weight BMI 18.5-24.9
* otorhinolaryngological surgeries

Exclusion Criteria:

* refusal to participate in the study;
* pregnancy or suspected pregnancy;
* neuromuscular diseases, renal or hepatic impairment;
* hepatic dysfunction;
* story or predictors of difficult airway;
* hypermagnesemia (Mg> 2.5 mEq / L);
* hypomagnesemia (Mg <1.7 mEq / L);
* furosemide, aminoglycosides, aminophylline azathioprine; cyclophosphamide, anti-inflammatory and magnesium;
* allergy to drugs used in the study;
* participants from other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of treatment with magnesium sulfate the T4 / T1 ratio . | 3 hours
  The T4 / T1 ratio after reversal with sugammadex deep and moderate neuromuscular blockade induced by rocuronium.Clinical tests and contraction of the adductor pollicis muscle in response to ulnar nerve train-of-four (TOF) stimulation was acceleromyographically quantified using a TOF-Watch SX.

SECONDARY OUTCOMES:
Record the possible serious respiratory events in the post-anesthetic recovery room | 1 hour after the end of surgery
  Obstruction of the upper airway that requires intervention; mild to moderate hypoxemia - lower saturation between 90% -93%, with no improvement after request to deep breathing or tactile stimulation; severe hypoxemia - saturation less than 90%, with no improvement after request to deep breathing or tactile stimulation; signs of increased work of breathing - more than 20 breaths per minute and use of accessory muscles; inability to breathe deeply when requested; via musculature of signs of weakness air higher, as speech disability; reintubation in the post anesthetic recovery room; clinical evidence or suspicion of bronchial aspiration after extubation (gastric contents oropharyngeal or tracheal tube accompanied by hypoxemia).
Evaluate the occurrence of any residual neuromuscular block in the post anesthetic recovery room | 1 hour after the end of surgery
  Clinical tests and contraction of the adductor pollicis muscle in response to ulnar nerve train-of-four (TOF) stimulation was acceleromyographically quantified using a TOF-Watch SX.
Record the evolution of the height of the first response (T1) | 1 hour after the end of surgery
  Clinical tests and contraction of the adductor pollicis muscle in response to ulnar nerve train-of-four (TOF) stimulation was acceleromyographically quantified using a TOF-Watch SX.
Record the possible occurrence of severe respiratory complications every 24 hours | 72 hours max
  Obstruction of the upper airway that requires intervention; mild to moderate hypoxemia - lower saturation between 90% -93%, with no improvement after request to deep breathing or tactile stimulation; severe hypoxemia - saturation less than 90%, with no improvement after request to deep breathing or tactile stimulation; signs of increased work of breathing - more than 20 breaths per minute and use of accessory muscles; inability to breathe deeply when requested; via musculature of signs of weakness air higher, as speech disability; reintubation in the post anesthetic recovery room; clinical evidence or suspicion of bronchial aspiration after extubation (gastric contents oropharyngeal or tracheal tube accompanied by hypoxemia).
Evaluate postoperative pain | 72 hours
  Use of visual analogue pain scale (0-10) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paulo A Germano Filho, MSc, Principal Investigator — Hospital Federal de Bonsucesso; Ismar L Cavalcanti, PhD, Study Director — Universidade Federal Fluminense; Nubia V Figueiredo, PhD, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Federal de Bonsucesso, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Unterbuchner C, Ziegleder R, Graf B, Metterlein T. Magnesium-induced recurarisation after reversal of rocuronium-induced neuromuscular block with sugammadex. Acta Anaesthesiol Scand. 2015 Apr;59(4):536-40. doi: 10.1111/aas.12461. Epub 2015 Jan 13. PMID 25582520
- [Result] Hans GA, Bosenge B, Bonhomme VL, Brichant JF, Venneman IM, Hans PC. Intravenous magnesium re-establishes neuromuscular block after spontaneous recovery from an intubating dose of rocuronium: a randomised controlled trial. Eur J Anaesthesiol. 2012 Feb;29(2):95-9. doi: 10.1097/EJA.0b013e32834e13a6. PMID 22183158
- [Result] Carron M, Ori C. Magnesium-induced recurarisation after reversal of rocuronium-induced neuromuscular block with sugammadex. Findings vs. speculation. Acta Anaesthesiol Scand. 2015 Aug;59(7):946-7. doi: 10.1111/aas.12551. Epub 2015 May 12. No abstract available. PMID 25962433